CLINICAL TRIAL: NCT01120223
Title: Safety and Efficacy of Calcipotriol Plus Betamethasone Dipropionate Gel in Adolescent Subjects (Aged 12 to 17) With Scalp Psoriasis
Brief Title: Safety and Efficacy of LEO 80185 Gel in Adolescent Subjects (Aged 12 to 17) With Scalp Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MBL 0412 INT; 2008-005456-24 (EudraCT Number)
Record Dates: First submitted 2010-04-09; First posted 2010-05-10 (Estimated); Results first posted 2014-12-01 (Estimated); Last update posted 2025-03-11 (Actual); Status verified 2015-03

CONDITIONS: Scalp Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LEO 80185 gel once daily application (Experimental)
  Interventions: Drug: LEO 80185 (Xamiol® gel/Taclonex® Scalp topical suspension)

INTERVENTIONS:
Drug: LEO 80185 (Xamiol® gel/Taclonex® Scalp topical suspension) — Once daily application

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of once daily use of LEO 80185 gel in adolescent subjects (aged 12 to 17) with scalp psoriasis. LEO 80185 gel has marketing approval in many countries under the brand names Xamiol® gel and Taclonex Scalp® Topical Suspension for the treatment of scalp psoriasis in adults. No studies have been performed in subjects younger than 18 years

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of scalp psoriasis which is of an extent of more than or equal to 10% of the scalp area
* A clinical diagnosis of scalp psoriasis which is of at least moderate severity according to the investigator's global assessment
* Serum albumin-corrected calcium below the upper reference limit at screening visit 2

Exclusion Criteria:

* A history of hypersensitivity to any component of the LEO 80185 gel
* Topical treatment on the trunk and/or limbs with very potent (WHO group IV) corticosteroids within 2 weeks prior to Visit 1 or during the study
* Topical treatment on the face and/or genital/skin folds with potent or very potent (WHO groups III-IV) corticosteroids within 2 weeks prior to Visit 1 or during the study
* Systemic treatment with biological therapies (marketed or not marketed), with a possible effect on scalp psoriasis within the following time period prior to Visit 1 and during the study:

  * etanercept - within 4 weeks prior to Visit 1
  * adalimumab, alefacept, infliximab - within 2 months prior to Visit 1
  * ustekinumab - within 4 months prior to Visit 1
  * experimental products - within 4 weeks/5 half-lives (whichever is longer) prior to Visit 1
* Systemic treatment with therapies other than biologicals, with a possible effect on scalp psoriasis (e.g., corticosteroids, retinoids, immunosuppressants, PUVA) within 4 weeks prior to Visit 1 (Day 0) or during the study
* UVB therapy within 2 weeks prior to Visit 1 or during the study
* Any topical treatment on the scalp (except for emollients and non-steroid medicated shampoos) within 2 weeks prior to Visit 1 or during the study
* Systemic calcium or vitamin D supplements, antacids, diuretics, antiepileptics, diphosphonates or calcitonin within 4 weeks prior to screening visit 2 or during the study
* Planned initiation of, or changes to, concomitant medication that could affect scalp psoriasis (e.g., betablockers, chloroquine, lithium, ACE inhibitors) during the study
* Current diagnosis of guttate, erythrodermic, exfoliative or pustular psoriasis
* Subjects with any of the following conditions present on the scalp area: viral (e.g., herpes or varicella) lesions of the skin, fungal and bacterial skin infections, parasitic infections, skin manifestations in relation to syphilis or tuberculosis, rosacea, acne vulgaris, acne rosacea, atrophic skin, striae atrophicae, fragility of skin veins, ichthyosis, ulcers and wounds
* Planned excessive exposure to sun during the study that may affect scalp psoriasis
* Known or suspected disorders of calcium metabolism associated with hypercalcaemia

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 78 (Actual)
Dates: Start 2010-05; Primary Completion 2012-08 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander V Anstey, MD, Principal Investigator — Royal Gwent Hospital
Locations (17):
- Canada (8):
  - Kirk Barber Research, Calgary, Alberta
  - Winnipeg Clinic Dermatology Research, Winnipeg, Manitoba
  - UltraNova Skincare, Barrie, Ontario
  - The Guenther Dermatology Research Centre, London, Ontario
  - Lynderm Research Inc., Markham, Ontario
  - SKiN Centre for Dermatology, Peterborough, Ontario
  - The Centre for Dermatology and Cosmetic Surgery, Richmond Hill, Ontario
  - Royal University Hospital, Division of Dermatology, Saskatoon, Saskatchewan
- CHU Saint-Etienne - Hôpital Nord, Service de Dermatologie, Saint-Etienne, France
- United Kingdom (8):
  - Monklands Hospital, Airdrie, Lanarkshire
  - Burbage Surgery, Burbage, Leicestershire
  - Whipps Cross University Hospital, Leytonstone, London
  - Hope Hospital, Salford, Manchester
  - Harrogate District Hospital, Harrogate, North Yorkshire
  - Leeds General Infirmary, Leeds, W. Yorkshire
  - City Hospital, Birmingham
  - Royal Gwent Hospital, Newport

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Trials at LEO Pharma — https://www.leopharmatrials.com/en

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Start date: 22-Nov-2010 Completion date: 15-Oct-2012
Pre-assignment Details: Prior to Visit 1 (Day 0), a wash-out period (up to 8 weeks, as defined by the exclusion criteria) was to be completed if the subject had been treated with antipsoriatic treatments or other relevant medication; 2 screening visits were planned.
Groups:
- LEO 80185 Gel Once Daily Application: Taclonex® Scalp Topical Suspension/Daivobet® gel /Dovobet® gel/Xamiol® gel Calcipotriol 50 mcg/g plus betamethasone 0.5 mg/g (as dipropionate) gel once daily for up to 8 week to treat psoriasis on the scalp.
Period: Overall Study
Arm/Group | LEO 80185 Gel Once Daily Application
Started | 78
Completed | 74
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | LEO 80185 Gel Once Daily Application
Number analyzed (Participants) | 78
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 78
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.6 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 35
Region of Enrollment [Number; unit: participants]
  France | 22
  Canada | 37
  United Kingdom | 19

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Adverse Drug Reactions (ADRs)
Description: Adverse events for which the investigator did not describe the causal relationship to IP as not related
Time Frame: Throughout trial, up to 8-weeks
Measure: Number; unit: percent subjects
Arm/Group | LEO 80185 Gel Once Daily Application
Number analyzed (Participants) | 78
percent subjects | 6.4

2. Primary Outcome: Change in Albumincorrected Serum Calcium From Baseline to Week 4
Description: Change in albumincorrected serum calcium from Baseline to week 4
Time Frame: Baseline and week 4
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | LEO 80185 Gel Once Daily Application
Number analyzed (Participants) | 77
mmol/L | -0.014 (0.139)

3. Primary Outcome: Change in Albumincorrected Serum Calcium From Baseline to Week 8
Description: Change in albumincorrected serum calcium from Baseline to week 8
Time Frame: Baseline and week 8
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | LEO 80185 Gel Once Daily Application
Number analyzed (Participants) | 60
mmol/L | -0.002 (0.098)

4. Secondary Outcome: Change in Plasma PTH From Baseline to Week 4
Description: Change in plasma PTH (parathyroid hormone) from Baseline to week 4
Time Frame: Baseline and week 4
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | LEO 80185 Gel Once Daily Application
Number analyzed (Participants) | 74
ng/L | 1.2 (16.0)

5. Secondary Outcome: Change in Plasma PTH From Baseline to Week 8
Description: Change in plasma PTH (parathyroid hormone) from Baseline to week 8
Time Frame: Baseline and week 8
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | LEO 80185 Gel Once Daily Application
Number analyzed (Participants) | 61
ng/L | -2.8 (13.0)

6. Secondary Outcome: Subjects With Controlled Disease (i.e., Clear or Almost Clear) According to the Investigator's Global Assessment (IGA) of Disease Severity at Week 2
Description: Disease severity of the scalp psoriasis as assessed by the 6-point scale IGA, based on the condition of the disease at the time of evaluation at week 2. The IGA Scale: 1 = clear, 2 = almost clear, 3 = mild, 4 = moderate, 5 = severe, and 6 = very severe.
Time Frame: Week 2
Measure: Number; unit: participants
Arm/Group | LEO 80185 Gel Once Daily Application
Number analyzed (Participants) | 78
participants | 37

7. Secondary Outcome: Subjects With Controlled Disease (i.e., Clear or Almost Clear) According to the Investigator's Global Assessment (IGA) of Disease Severity at Week 4
Description: Disease severity of the scalp psoriasis as assessed by the 6-point scale IGA, based on the condition of the disease at the time of evaluation at week 4
Time Frame: Week 4
Measure: Number; unit: participants
Arm/Group | LEO 80185 Gel Once Daily Application
Number analyzed (Participants) | 78
participants | 59

8. Secondary Outcome: Subjects With Controlled Disease (i.e., Clear or Almost Clear) According to the Investigator's Global Assessment (IGA) of Disease Severity at Week 8
Description: Disease severity of the scalp psoriasis as assessed by the 6-point scale IGA, based on the condition of the disease at the time of evaluation at week 8
Time Frame: Week 8
Measure: Number; unit: participants
Arm/Group | LEO 80185 Gel Once Daily Application
Number analyzed (Participants) | 61
participants | 49

9. Primary Outcome: Change in Albumincorrected Serum Calcium From Baseline to End of Treatment
Description: Change in albumincorrected serum calcium from Baseline to end of treatment
Time Frame: Baseline and End of treatment (up to 8 weeks)
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | LEO 80185 Gel Once Daily Application
Number analyzed (Participants) | 78
mmol/L | 0.000 (0.101)

10. Primary Outcome: Change in 24-hour Urinary Calcium Excretion From Baseline to Week 4
Description: Change in 24-hour urinary calcium excretion from Baseline to week 4
Time Frame: Baseline and week 4
Measure: Mean (Standard Deviation); unit: mmol/24hr
Arm/Group | LEO 80185 Gel Once Daily Application
Number analyzed (Participants) | 76
mmol/24hr | -0.01 (1.54)

11. Primary Outcome: Change in 24-hour Urinary Calcium Excretion From Baseline to Week 8
Description: Change in 24-hour urinary calcium excretion from Baseline to week 8
Time Frame: Baseline and week 8
Measure: Mean (Standard Deviation); unit: mmol/24hr
Arm/Group | LEO 80185 Gel Once Daily Application
Number analyzed (Participants) | 60
mmol/24hr | 0.03 (1.42)

12. Primary Outcome: Change in 24-hour Urinary Calcium Excretion From Baseline to End of Treatment
Description: Change in 24-hour urinary calcium excretion from Baseline to end of treatment
Time Frame: Baseline and End of treatment (up to 8 weeks)
Measure: Mean (Standard Deviation); unit: mmol/24hr
Arm/Group | LEO 80185 Gel Once Daily Application
Number analyzed (Participants) | 77
mmol/24hr | -0.03 (1.43)

13. Primary Outcome: Change in Urinary Calcium:Creatinine Ratio From Baseline to Week 4
Description: Change in urinary calcium:creatinine ratio from Baseline to week 4
Time Frame: Baseline and week 4
Measure: Mean (Standard Deviation); unit: mmol/g
Arm/Group | LEO 80185 Gel Once Daily Application
Number analyzed (Participants) | 76
mmol/g | -0.269 (1.684)

14. Primary Outcome: Change in Urinary Calcium:Creatinine Ratio From Baseline to Week 8
Description: Change in urinary calcium:creatinine ratio from Baseline to week 8
Time Frame: Baseline and week 8
Measure: Mean (Standard Deviation); unit: mmol/g
Arm/Group | LEO 80185 Gel Once Daily Application
Number analyzed (Participants) | 60
mmol/g | -0.003 (1.500)

15. Primary Outcome: Change in Urinary Calcium:Creatinine Ratio From Baseline to End of Treatment
Description: Change in urinary calcium:creatinine ratio from Baseline to end of treatment
Time Frame: Baseline and End of treatment (up to 8 weeks)
Measure: Mean (Standard Deviation); unit: mmol/g
Arm/Group | LEO 80185 Gel Once Daily Application
Number analyzed (Participants) | 77
mmol/g | -0.1156 (1.679)

16. Secondary Outcome: Subjects With Controlled Disease (i.e., Clear or Almost Clear) According to the Investigator's Global Assessment (IGA) of Disease Severity at End of Treatment
Description: Disease severity of the scalp psoriasis as assessed by the 6-point scale IGA, based on the condition of the disease at the time of evaluation at end of treatment
Time Frame: End of treatment (up to 8 weeks)
Measure: Number; unit: participants
Arm/Group | LEO 80185 Gel Once Daily Application
Number analyzed (Participants) | 78
participants | 66

17. Secondary Outcome: Percentage Change in Total Sign Score (TSS; Sum of Severity Scores for Each Individual Clinical Sign, Redness, Thickness, and Scaliness)From Baseline to Week 2
Description: Investigator assessment of scalp psoriasis lesions in terms of the three clinical signs: redness, thickness, and scaliness. Each clinical sign, a single score (ranging from 0 to 4), reflecting the average severity of all psoriatic lesions on the scalp, were determined. The sum of the three scores (redness, thickness, and scaliness) constitutes the Total Sign Score of the psoriasis on scalp, ranging from 0 (best possible outcome) to 12 points (worst possible outcome).
Time Frame: Baseline and week 2
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | LEO 80185 Gel Once Daily Application
Number analyzed (Participants) | 78
percentage of change | -62.7 (22.3)

18. Secondary Outcome: Percentage Change in Total Sign Score (TSS; Sum of Severity Scores for Each Individual Clinical Sign, Redness, Thickness, and Scaliness) From Baseline to Weeks 4
Description: Investigator assessment of scalp psoriasis lesions in terms of the three clinical signs: redness, thickness, and scaliness. Each clinical sign, a single score (ranging from 0 to 4), reflecting the average severity of all psoriatic lesions on the scalp, were determined. The sum of the three scores (redness, thickness, and scaliness) constitutes the Total Sign Score of the psoriasis on scalp, ranging from 0 to 12 points.
Time Frame: Baseline and week 4
Measure: Mean (Standard Deviation); unit: percent of change
Arm/Group | LEO 80185 Gel Once Daily Application
Number analyzed (Participants) | 78
percent of change | -72.1 (21.4)

19. Secondary Outcome: Percentage Change in Total Sign Score (TSS; Sum of Severity Scores for Each Individual Clinical Sign, Redness, Thickness, and Scaliness) From Baseline to Week 8
Description: as for outcome 17
Time Frame: Baseline and week 8
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | LEO 80185 Gel Once Daily Application
Number analyzed (Participants) | 61
percent change | -76.6 (23.5)

20. Secondary Outcome: Percentage Change in Total Sign Score (TSS; Sum of Severity Scores for Each Individual Clinical Sign, Redness, Thickness, and Scaliness) From Baseline to End of Treatment.
Description: as for outcome 17
Time Frame: Baseline and End of treatment (up to 8 weeks)
Measure: Mean (Standard Deviation); unit: percent of change
Arm/Group | LEO 80185 Gel Once Daily Application
Number analyzed (Participants) | 78
percent of change | -80.4 (22.6)

21. Secondary Outcome: Subjects With Controlled Disease (Defined as Clear or Very Mild) According to the Patient's Global Assessment of Disease Severity at Week 2
Description: Disease severity of the scalp psoriasis as assessed by the 5-point scale, Patient's Global Assessment of Disease Severity, based on the condition of the disease at the time of evaluation. The scale: 1 = clear, 2 = very mild, 3 = mild, 4 = moderate, 5 = severe.
Time Frame: Week 2
Measure: Number; unit: participants
Arm/Group | LEO 80185 Gel Once Daily Application
Number analyzed (Participants) | 78
participants | 44

22. Secondary Outcome: Subjects With Controlled Disease (Defined as Clear or Very Mild) According to the Patient's Global Assessment of Disease Severity at Week 4
Description: Disease severity of the scalp psoriasis as assessed by the 5-point scale, Patient's Global Assessment of Disease Severity, based on the condition of the disease at the time of evaluation.
Time Frame: Week 4
Measure: Number; unit: participants
Arm/Group | LEO 80185 Gel Once Daily Application
Number analyzed (Participants) | 78
participants | 55

23. Secondary Outcome: Subjects With Controlled Disease (Defined as Clear or Very Mild) According to the Patient's Global Assessment of Disease Severity at Week 8
Description: as for outcome 22
Time Frame: Week 8
Measure: Number; unit: participants
Arm/Group | LEO 80185 Gel Once Daily Application
Number analyzed (Participants) | 61
participants | 51

24. Secondary Outcome: Subjects With Controlled Disease (Defined as Clear or Very Mild) According to the Patient's Global Assessment of Disease Severity at End of Treatment
Description: as for outcome 22
Time Frame: End of treatment (up to 8 weeks)
Measure: Number; unit: participants
Arm/Group | LEO 80185 Gel Once Daily Application
Number analyzed (Participants) | 78
participants | 68

25. Secondary Outcome: Withdrawal
Description: How many subjects withdrew from the study. Reasons for withdrawal:
  due to exclusion criteria emerging, due to AE(s), or due to other reason
Time Frame: Week 4 and 8
Measure: Number; unit: participants
Arm/Group | LEO 80185 Gel Once Daily Application
Number analyzed (Participants) | 78
participants | 4

ADVERSE EVENTS:
Arm/Group | LEO 80185 Gel Once Daily Application
Serious Adverse Events (participants affected / at risk) | 0/78
Other Adverse Events (participants affected / at risk) | 10/78
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LEO 80185 Gel Once Daily Application (N=78)
Headache (Nervous system disorders) | 4
Pharyngitis (Infections and infestations) | 4
Upper respiratory tract infection (Infections and infestations) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
LEO acknowledges the investigators' right to publish the results of the trial, irrespective of outcome. Pubs/presentations by investigator(s) shall not be made before the results of a joint publication is public. LEO retains the right to have any publication submitted to LEO for review at least 30 days prior to this paper being submitted for publication/presentation. Investigators must undertake not to submit any part of their individual data for publication without the prior consent of LEO.